CLINICAL TRIAL: NCT03231878
Title: A Randomized, Double-blind, Placebo-controlled, Multinational, Multicenter Study With Open-label Treatment Extension to Assess the Effect of MIN-102 (IMP) on the Progression of Adrenomyeloneuropathy in Male Patients With X-linked Adrenoleukodystrophy
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of MIN-102 (IMP) in Male AMN Patients.
Acronym: Advance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Minoryx Therapeutics, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-2-01
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Adrenoleukodystrophy
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: MIN-102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: MIN-102 — MIN-102 treatment
  Arms: Active
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II/III, randomized, double-blind, placebo-controlled, multicenter, two parallel-group study in male patients with the AMN phenotype of X-linked adrenoleukodystrophy (X-ALD) to assess the efficacy and safety of MIN-102 treatment. Study sites will consist of specialist referral centers experienced in the management of adrenoleukodystrophy (ALD).

ELIGIBILITY:
Inclusion Criteria:

* Male and between 18-65 years of age.
* Diagnosed with X-linked adrenoleukodystrophy (X-ALD) based on elevated VLCFA and genetic testing.
* Clinical evidence of spinal cord involvement.

Exclusion Criteria:

* Any other chronic neurological disease with signs of spastic paraplegia, such as hereditary spastic paraplegia, multiple sclerosis, etc.
* Presence of inflammatory (Gd-enhancing) MRI lesions or any abnormality other than those mentioned in the inclusion criteria.
* Known type 1 or type 2 diabetes.
* Known intolerance to pioglitazone or any other thiazolidinedione.
* Taking or have taken honokiol, pioglitazone or other thiazolidinediones within the 6 months prior to screening.
* Previous bone marrow transplantation.
* Previous or current history of cancer (other than treated basal cell carcinoma).
* Previous or current history of congestive heart failure.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of MIN-102 on the progression of adrenomyeloneuropathy (AMN) in male patients as determined by a motor function test. | in 96 weeks

SECONDARY OUTCOMES:
To evaluate the efficacy of MIN-102 in terms of patient reported outcomes. | in 96 weeks
SSPROM (Severity Score System for Progressive Myelopathy ) | in 96 weeks
EDSS (Expanded Disability Status Scale ) | in 96 weeks
Quality of life scales (Euroqol) | in 96 weeks
Incidence of cerebral inflammatory lesions | in 96 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
- Hospital de la Pitié-Salpêtrière, Paris, France
- Universitat Leipzig Klinik and Poliklinik für Neurologie, Leipzig, Germany
- Institute of Genomic Medicine and Rare Disorders, Budapest, Hungary
- Instituto Neurologico Carlo Besta, Milan, Italy
- Academish Medisch Centrum, Amsterdam, Netherlands
- Hospital Universitari Vall d'Hebrón, Barcelona, Spain
- National hospital for Neurology and Neurosurgery Charles Dent Metabolic Unit), London, United Kingdom

REFERENCES:
- [Derived] Kohler W, Engelen M, Eichler F, Lachmann R, Fatemi A, Sampson J, Salsano E, Gamez J, Molnar MJ, Pascual S, Rovira M, Vila A, Pina G, Martin-Ugarte I, Mantilla A, Pizcueta P, Rodriguez-Pascau L, Traver E, Vilalta A, Pascual M, Martinell M, Meya U, Mochel F; ADVANCE Study Group. Safety and efficacy of leriglitazone for preventing disease progression in men with adrenomyeloneuropathy (ADVANCE): a randomised, double-blind, multi-centre, placebo-controlled phase 2-3 trial. Lancet Neurol. 2023 Feb;22(2):127-136. doi: 10.1016/S1474-4422(22)00495-1. PMID 36681445